CLINICAL TRIAL: NCT06911762
Title: The Effects of a Structured Hand Exercise Program on Trigger Finger: A Randomized Controlled Trial
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Hong Kong Polytechnic University (Other)
Responsible Party: Principal Investigator, Freddy Man Hin LAM, Assistant Professor, The Hong Kong Polytechnic University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HSEARS20241227004
Record Dates: First submitted 2025-03-28; First posted 2025-04-04 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2025-03

CONDITIONS: Trigger Finger
Keywords: Trigger finger; tenosynovitis; physiotherapy; conservative treatment; Exercise
MeSH Terms: conditions — Trigger Finger Disorder; Tenosynovitis; Motor Activity | interventions — Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Exercise (Experimental)
  Interventions: Behavioral: Exercise
- Control (No Intervention): Participants will receive no intervention.

INTERVENTIONS:
Behavioral: Exercise — Participants will receive a 6-week structured hand exercise program. Participants will attend a face-to-face exercise session to learn all hand exercises. The exercise program will include: (1) Finger flexor stretching, (2) Tendon gliding exercise and (3) Isometric finger flexor exercise. A weekly tele follow-up will be done to participants in the experimental group
  Arms: Exercise

SUMMARY:
To explore the effectiveness of a structured hand exercise program as a conservative treatment for trigger finger.

ELIGIBILITY:
Inclusion Criteria:

* Adults with aged > 18 years old who are diagnosed with trigger finger
* The Green classification grade 2 or grade 3
* Pain (NPRS) equal or more than 4/10, during active triggering

Exclusion Criteria:

* Pediatric or congenital trigger finger
* Previously received physiotherapy, corticosteroid injection or surgery for trigger finger
* Hand trauma, local infection or using systemic steroids due to other diseases

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Estimated)
Dates: Start 2025-04-15 (Estimated); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-08-01 (Estimated)

PRIMARY OUTCOMES:
Numeric Pain Rating Scale (NPRS) during triggering or movement | Baseline, 6 weeks after baseline, 10 weeks after baseline
  NPRS consists of 11-point numeric scale from '0' (no pain) to '10' (worst pain imaginable). Participants rate the pain level based on their own pain intensity from 0-10

SECONDARY OUTCOMES:
Trigger finger stage in the Green Classification | Baseline, 6 weeks after baseline, 10 weeks after baseline
  Green's classification for trigger finger: Grade 1 (A history of catching with local pain). Grade 2 (Demonstrable catching with normal active extension). Grade 3 (Demonstrable locking requiring passive extension). Grade 4 (Fixed flexion deformity)
Frequency of triggering | Baseline, 6 weeks after baseline, 10 weeks after baseline
  The frequency of triggering will be represented by the number of triggering events in ten active fists, from 0 to 10. Two questions will be asked: (1) What is the average number of triggering in ten active fists in the past one week? (2) What is the average number of painful triggering in ten active fists in the past one week?
Functional score by Quick Disabilities of the Arm, Shoulder, and Hand Questionnaire (Hong Kong version) | Baseline, 6 weeks after baseline, 10 weeks after baseline
  Quick Disabilities of the Arm, Shoulder, and Hand Questionnaire (QuickDASH) is a shorten version of the Disabilities of the Arm, Shoulder, and Hand Questionnaire (DASH). QuickDASH consisted of 11 items to measure physical function and symptoms in patients with upper limb disorders. DASH and QuickDASH were translated into Hong Kong version. Participants must complete at least 10 of the 11 items for a score to be calculated and the scores range from 0 (no disability) to 100 (most severe disability).
Grip strength of the affected hand | Baseline, 6 weeks after baseline, 10 weeks after baseline
  Grip strength will be assessed using the American Society of Hand Therapists (ASHT) protocol. Participants will be seated in a chair without arm rests, with hips and knees in 90 degrees. Shoulder holds in adduction and neutral rotation. Elbow holds in 90 degrees flexion with forearm in neutral rotation. Participants grip the dynamometer in 15-30 degrees wrist extension and 0-15 degrees of ulnar deviation. Participants will be asked to grip the dynamometer as hard as they can for 3 trials. The mean of the 3 trials will be recorded as the grip strength in kg.
Structural changes using musculoskeletal ultrasound (A1 pulley thickness, flexor tendon thicknesses, A1 pulley lumen size) | Baseline, 6 weeks after baseline, 10 weeks after baseline
  Musculoskeletal ultrasound with a linear transducer (12MHz probe) will be used to evaluate the structural outcome measures.

CONTACTS AND LOCATIONS:
Locations (1):
- The Hong Kong Polytechnic University, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: Yes
The study data can be provided via contacting the Principal Investigator
Supporting Information: Study Protocol, SAP, ICF, CSR